CLINICAL TRIAL: NCT04973904
Title: A Single-Arm, Multicenter, Phase II Study to Investigate Efficacy and Safety of Toripalimab Combined With Chemotherapy and Bevacizumab as First-Line Treatment in Patients With Recurrent, Refractory and Metastatic Cervical Cancer
Brief Title: Toripalimab Combined With Chemotherapy and Bevacizumab as First-Line Treatment in Patients With Advanced Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-ISS-CO214
Record Dates: First submitted 2021-07-08; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Cervical Cancer
Keywords: Toripalimab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — toripalimab; Paclitaxel; Cisplatin; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1+Paclitaxel+Cisplatin+Bevacizumab (Experimental): Toripalimab 240mg intravenously(IV) every 3 weeks (Q3W)
  Paclitaxel 175mg/m2 IV every 3 weeks (Q3W)
  Cisplatin 50mg/m2 (Q3W)
  Bevacizumab 7.5mg/kg IV every 3 weeks (Q3W)
  Interventions: Drug: Toripalimab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Toripalimab — IV infusion
Drug: Paclitaxel — IV infusion
Drug: Cisplatin — IV infusion
Drug: Bevacizumab — IV infusion

SUMMARY:
This is a single-arm, multicenter, phase II study to investigate efficacy and safety of Toripalimab combined with chemotherapy (paclitaxel and cisplatin) and Bevacizumab as first-line treatment in patients with recurrent, refractory and metastatic cervical cancer

DETAILED DESCRIPTION:
The objective of this study is to evaluate the efficacy and safety of therapy with toripalimab andchemotherapy (paclitaxel and cisplatin) and Bevacizumab as first-line treatment in patients with recurrent, refractory and metastatic cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Cervical squamous cell carcinoma, adenocarcinoma and adenosquamous cell carcinoma diagnosed by histopathology
* FIGO stage IVB according to 2018 FIGO staging classification; Any FIGO stage with persistent or progressed lesions after treatment; Any FIGO stage with recurrent lesions and recurrent-free interval > 6 month
* Subjects has not been treated with systemic chemotherapy and is not amenable to curative treatment (such as with surgery and/or radiation). Subject who previously treated with cisplatin-based CCRT is allowed
* Has measurable disease per RECIST 1.1
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Written and signed informed consent.
* Patients must have adequate function as defined:

  1. ANC≥1.5*10^9/L; PLT≥100*10^9/L, Hb≥90 g/L, WBC≥3.5*10^9/L
  2. Total Bilirubin (TBIL)≤1.5*Upper Limit of Normal(UNL)
  3. Alanine Transaminase (ALT)and Aspartate Aminotransferase(AST)≤2.5*ULN.For liver metastasis patients, ALT and AST≤5*ULN, Alkaline phosphatase (ALP) ≤ 3 x UNL. For liver metastasis patients, Alkaline phosphatase (ALP) ≤ 5 x UNL
  4. Cr≤ ULN, or creatinine clearance rate ≥60 mL/min,
* Proteinuria ≤1+，if proteinuria≥ 1+ and 24 hours total urine protein ≤ 1.0 g
* Patients who did not receive anticoagulant therapy: INR ≤ 1.5 × ULN. If the patient receives prophylactic anticoagulant therapy, the INR ≤ 2 × ULN within 14 days before the start of the study treatment and the activated partial thromboplastin time is within the normal range, acceptable for enrollment
* Has not a history of autoimmune diseases
* Controlled hepatitis B or hepatitis C subjects are eligible to participate in the study as long as they meet the following criteria: The HBV viral load must be less than 2,000 IU/mL (< 10000 copies/ml). Subjects have received anti-HBV therapy for 2 weeks before starting the study treatment and should maintain the same treatment throughout the study treatment period. Subjects with positive HCV RNA should receive anti-HCV therapy and liver function ≤ CTCAE Grade 1.
* Subjects has not received corticosteroids or other immunosuppressive medications within 14 days prior to the study treatment.
* Female subjects must not be pregnant, not breastfeeding, and at least one of the following conditions can be included in the study: women who do not have fertility or who agree to be at least 60 days after the treatment and the last study drug administration Fertility women who take contraceptive measures as required by the programme.

Exclusion Criteria:

* Prior systemic treatment for recurrent, secondarily progressive or initially metastatic disease
* Indications for potentially curative treatment (surgery or radiation therapy)
* Has received prior radiotherapy within 2 weeks before enrollment,or has not recovered from the effects of radiotherapy.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with known brain metastases may participate provided that the brain metastases have been previously treated with radiotherapy or surgery only and are radiographically stable
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once a month or more frequently); Patients with stable symptoms for at least two weeks after drainage could be enrolled
* Patients with cirrhosis of any cause
* Major surgery, open biopsy or major trauma were performed within 28 days before the first dose of treatment
* Gastrointestinal or other active bleeding, gastrointestinal perforation
* History of organ fistula (such as gallbladder fistula, tracheal fistula, pancreatic fistula, etc.)
* Coagulation disorder or thromboembolic disease without standard anticoagulant therapy
* uncontrolled hypertension, hypertensive crisis, hypertensive encephalopathy
* Patients with severe wounds that cannot be healed, ulcers or fractures
* Grade ≥ 3 venous thromboembolic events (VTE)
* History of arterial thromboembolism
* Acute intestinal obstruction in the last 6 months
* A history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months
* Previous use of any anti-PD-1, anti-PD-L1 / L2 antibody, anti-CTLA-4 antibody and other immunotherapy and VEGF/VEGFR inhibitors (including bevacizumab)
* Known hypersensitivity or allergy to paclitaxel, cisplatin, carboplatin, bevacizumab, Toripalimab or any of their excipients.
* Another malignant tumor is known and is currently undergoing progress or has been actively treated in the past 3 years. Note: Subjects who have received skin basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ (eg, breast cancer, bladder cancer in situ) that may be curable may be treated.
* Major surgery was performed within 3 weeks before enrollment or had not completely recovered from the previous surgery (the definition of major surgery refers to the level 3 and level 4 surgery in the administrative measures for clinical application of medical technology implemented on May 1, 2009)
* Known mental illness or substance abuse conditions can impede the ability of the subject to meet research requirements
* Poor compliance
* Active pulmonary tuberculosis (TB), who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within one year before the first dose of treatment
* A history of positive HIV
* Patients with acute or chronic hepatitis B or hepatitis C infection, HBV DNA > 2000 IU / ml or 104 copies / ml; HCV RNA > 103 copies / ml; Hepatitis B surface antigen (HbsAg) and anti HCV antibody double positive.
* Active autoimmune diseases, or have a history of autoimmune diseases or syndrome requiring systemic steroid / immunosuppressant use, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism, hypothyroidism, etc
* Administration of a live, attenuated vaccine within 28 days before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study
* Currently participating in other clinical trials
* Serious and uncontrollable comorbidities that may affect the compliance of the protocol or interfere with the results, including active opportunistic infections or advanced (severe) infections, uncontrolled diabetes, cardiovascular diseases (grade III or IV heart failure defined by the New York Heart Association classification), cardiac conduction block > secondary degree, myocardial infarction in the past 6 months, Unstable arrhythmia or unstable angina pectoris, cerebral infarction within 3 months, etc.) or pulmonary diseases (history of interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm)
* Pregnant or lactating women
* A history of allogeneic stem cell transplantation or organ transplantation
* Patients who were not suitable for this study due to other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) using RECIST v1.1

SECONDARY OUTCOMES:
Disease control rate | 1 year
  The proportion of patients with at least one tumor scan of complete response (CR) or partial response (PR) or stable disease (SD) using RECIST v1.1.
progression free survival | 3 years
  Time from cycle 1, day 1 of treatment to disease progression or death due to any cause
Overall survival | 3 years
  Time from cycle 1, day 1 of treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li C, Liu S, He Y, Yao H, Yuan Z, Yang J, Cao D, Cheng N, Yang J, Peng P, Xiang Y. Toripalimab combined with bevacizumab plus chemotherapy as first-line treatment for refractory recurrent or metastatic cervical cancer: a single-arm, open-label, phase II study (JS001-ISS-CO214). J Gynecol Oncol. 2025 May;36(3):e44. doi: 10.3802/jgo.2025.36.e44. Epub 2024 Oct 25. PMID 39482930